CLINICAL TRIAL: NCT04374383
Title: Clinical Effects of a Single Application of a Novel Photosensitizer in The Treatment of Chronic Periodontitis - A Randomized Controlled Trial
Brief Title: Novel Photosensitizer in The Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/2/2019
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis; Alveolar Bone Loss
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- main treatment group (Experimental): LASER assisted SRP followed by antimicrobial photodynamic therapy with a novel photosensitizer dye Phthalocyanine
  Interventions: Drug: Phthalocyanine Dye; Drug: LASER assisted SRP
- control group (Placebo Comparator): LASER assisted SRP
  Interventions: Drug: LASER assisted SRP

INTERVENTIONS:
Drug: Phthalocyanine Dye — following LASER assisted SRP, a novel photosensitizer phthalocyanine dye will be placed
  Other Names: Experimental group
  Arms: main treatment group
Drug: LASER assisted SRP — LASER assisted SRP will be carried
  Other Names: Control group

SUMMARY:
The aim of this study is to evaluate the periodontal outcomes after applying antimicrobial photodynamic therapy with a novel photosensitizer as compared to LASER assisted scaling and root planing alone.

DETAILED DESCRIPTION:
LASER assisted SRP followed by antimicrobial photodynamic therapy with a novel photosensitizer dye Phthalocyanine will be done in test group subjects.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients of age 30-60 years with generalized probing pocket depths (PPD) indicative of chronic periodontitis and with atleast two sites with PPD ≥5mm in each quadrant

Exclusion Criteria:

* Medically compromised patients, Subjects with a history of periodontal intervention within 6 months of the commencement of the study and smokers

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Release profile of the drug | Change from baseline to 7-days.
  Release profile of the drug in Gingival Crevicular Fluid (GCF) samples will be evaluated through biochemical testing kits.
probing pocket depths (PPD) | Change from baseline to 6-months.
  Assessment of probing pocket depths (PPD, in mm) by using a manual periodontal probe on six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual and distolingual) will be performed.
clinical attachment level (CAL) | Change from baseline to 6-months.
  Assessment of clinical attachment level (CAL, in mm) by using a manual periodontal probe on six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual and distolingual) will be performed.

SECONDARY OUTCOMES:
plaque index (PI) | Change from baseline to 6-months.
  Assessment of plaque (PI) - according to Turesky modification of Quigley and Hein Plaque Index; 0-No plaque 1-Isolated flecks of plaque at the gingival margin 2-A continuous band of plaque up to 1mm at the gingival margin 3-Plaque greater than 1mm in width and covering up to one third of the tooth surface 4-Plaque covering from one thirds to two thirds of the tooth surface 5-Plaque covering more than two thirds of the tooth surface.
bleeding on probing (BOP) | Change from baseline to 6-months.
  Assessment of bleeding on probing (BOP) as a dichotomous variable ("Yes"/"No") by using a manual periodontal probe.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - R V Chandra, Hyderabad, Telangana
  - SVS Institute of Dental Sciences, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No